CLINICAL TRIAL: NCT02516995
Title: Functional Magnetic Resonance Imaging for High Throughput Curietherapy Planning in Prostate Cancer
Acronym: FIBROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A00440-39; 2010/1630 (Other: CSET number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-06 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with prostate cancer (Experimental)
  Interventions: Device: Functional magnetic resonance imaging; Device: Ultrasound

INTERVENTIONS:
Device: Functional magnetic resonance imaging
Device: Ultrasound

SUMMARY:
Merge the data of ultrasound with that of the anatomical and functional MRI is necessary since the high dose rate Curietherapy is carried out under ultrasound guidance. The investigators will recruit prostate cancer patients to evaluate the quality of the data, their sensitivity to exam conditions (patient position, volume of endorectal probe, gold grains implanted before intensity modulated radiotherapy , IMRT) and to merge data from different sources with the purpose of estimating the opportunities of integration treatment plan for Curietherapy broadband.

The nuclear magnetic resonance imaging provides precise anatomical study, but also provides access to a functional approach to the tumor mapping of water diffusion coefficient (DW-MRI), for dynamic imaging with injection contrast agent (DCE-MRI) and finally by spectroscopic imaging (IRMS). This multimodality imaging project is part of a multidisciplinary context, involving close collaboration between clinicians, medical physicists, and physicists of the teams participating in this project (Institut Gustave Roussy and U2R2M-CIERM hospital Kremlin-Bicetre).

ELIGIBILITY:
Inclusion Criteria:

Patients with prostate cancer biopsy-proven, intermediate or high risk (according to D'Amico Classification), for which radiotherapy is indicated.

* Accepting the imaging tests.
* Age <70 years.
* Informed consent signed.

Exclusion Criteria:

* Mental pathology that can interfere with the proper conduct of the study;
* Claustrophobia;
* Severe heart or respiratory disorder that can make it difficult to achieve relatively long imaging tests
* Contraindications to magnetic resonance imaging (MRI)

  1. pacemaker, other electronic appliance (depending on model);
  2. heart valve, intra-cranial clip aneurysm, cerebral ventricular bypass valve (depending on model);
  3. intraocular metallic foreign bodies (chips), and other locations, according to the site to discuss.
  4. metal tracheostomy cannula;
  5. endovascular stent or vascular embolization coils placed within six weeks in advance;
  6. the impediments to a long examination with spectroscopy sequence of ten to twenty minutes: major tremors, inability to lie more than 30 minutes;
  7. local sources of magnetic distortion which is sensitive spectroscopic imaging: hip replacement, prostate biopsy older than six weeks.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quality of imaging [good/good enough/not good enough] | Assessed six weeks after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France